CLINICAL TRIAL: NCT05906524
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of KD6001 in Combination With Tislelizumab±Bevacizumab in Patients With Advanced HCC and Other Solid Tumors
Brief Title: KD6001 in Combination With Anti-PD-1 Antibody±Bevacizumab in Patients With Advanced HCC and Other Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Kanda Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KD6001CT03
Record Dates: First submitted 2023-05-24; First posted 2023-06-18 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-05

CONDITIONS: Advanced HCC; Other Solid Tumors
MeSH Terms: interventions — tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1：KD6001+Tislelizumab (Experimental): KD6001 combined with Tislelizumab in patients with solid tumors（hepatocellular carcinoma, esophageal squamous cell carcinoma, MSI-H or dMMR solid tumors are preferentially included）
  Interventions: Drug: KD6001; Drug: Tislelizumab
- Phase 2：KD6001+Tislelizumab±Bevacizumab (Experimental): KD6001 combined with Tislelizumab±Bevacizumab in patients with advanced HCC
  Interventions: Drug: KD6001; Drug: Tislelizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: KD6001 — KD6001 will be administered intravenously.
Drug: Tislelizumab — Tislelizumab will be administered intravenously.
Drug: Bevacizumab — Bevacizumab will be administered intravenously.
  Arms: Phase 2：KD6001+Tislelizumab±Bevacizumab

SUMMARY:
This is a phase 1b/2, open label study to evaluate the safety, tolerability, pharmacokinetics and initial efficacy of KD6001 in combination with Tislelizumab ± Bevacizumab in patients with Advanced HCC and Other Solid Tumors.

ELIGIBILITY:
Main Inclusion Criteria:

1. Being voluntary to sign the informed consent form.
2. Male or female, aged ≥ 18 years.
3. Patients whose estimated survival time is more than 3 months.
4. Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1.
5. At least one measurable lesion is used as the target lesion according to the Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST V1.1).
6. Histologically or cytologically confirmed advanced solid tumors. Have a current liver function meeting Child Pugh Class A in patients with HCC.

   Part A: Advanced solid tumors. PartB/C: HCC.
7. Patients will agree to provide tumor tissue samples.
8. The results of laboratory examination during the screening period suggest that the subjects have good organ function.
9. Male subjects with reproductive ability or female subjects with the possibility of pregnancy use effective contraceptive methods.
10. Good compliance and follow-up.

Main Exclusion Criteria:

1. History of malignancy other than the disease under study within 5 years prior to screening，except those malignancies that are expected to be cured after treatment.
2. Systematic treatment with antitumor drugs within 4 weeks prior to the start of this study.
3. Prior treatment with anti-CTLA-4 antibody.
4. Adverse events caused by prior treatment did not recovered to NCI-CTCAE v5.0 grade 1 and below.
5. Subjects with CNS metastases or leptomeningeal disease.
6. Subjects with an active, known or suspected autoimmune disease.
7. Subjects with acute or chronic active hepatitis B or hepatitis C.
8. Has histological or cytological diagnosis of fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma.
9. Subjects suffers from severe cardiovascular and cerebrovascular diseases. History or evidence of bleeding diathesis or significant coagulopathy at risk of bleeding.
10. Subjects with an active infection requiring systemic treatment.
11. Known history of testing positive for human immunodeficiency virus (HIV).
12. Subjects known to have active tuberculosis (TB).
13. Pregnant or breastfeeding females.
14. Known to be allergic to KD6001, tislelizumab, bevacizumab or its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to Day 21
  DLTs will be assessed during the dose-escalation phase and are defined as the following treatment-related adverse events occurring within a total of 21 days after the first trial administration.
The incidence and safety profile of participants with adverse events (AEs), serious adverse events(SAE), and immune-related adverse event(irAE) | Baseline to study completion up to 2 years
  Evaluate the adverse events (AE) according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 (NCI CTCAE 5.0).

SECONDARY OUTCOMES:
The antitumor activity of KD6001 in combination with Tislelizumab ± Bevacizumab measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Baseline to study completion up to 2 years
  Number of participants with response according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
Maximum Plasma Concentration [Cmax] | Baseline to study completion up to 2 years
  The PK profile of KD6001 in combination with Tislelizumab ± Bevacizumab.
Time to reach maximum serum concentration (Tmax) | Baseline to study completion up to 2 years
  The PK profile of KD6001 in combination with Tislelizumab ± Bevacizumab.
Half-life (T1/2) | Baseline to study completion up to 2 years
  The PK profile of KD6001 in combination with Tislelizumab ± Bevacizumab.
Area under blood concentration-time curve(AUC0-T and AUC0-∞) | Baseline to study completion up to 2 years
  The PK profile of KD6001 in combination with Tislelizumab ± Bevacizumab.
Apparent volume of distribution (Vd) | Baseline to study completion up to 2 years
  The PK profile of KD6001 in combination with Tislelizumab ± Bevacizumab.
The immunogenicity of KD6001 in combination with Tislelizumab ± Bevacizumab | Baseline to study completion up to 2 years
  Including the incidence of ADA positive. For ADA positive patients, the incidence of neutralizing antibody (Nab) will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, China